CLINICAL TRIAL: NCT02761564
Title: Restrictive Transfusion Strategy Early After Cardiac Surgery
Brief Title: SvO2 Trigger in Transfusion Strategy After Cardiac Surgery
Acronym: ReTSEACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 9655
Record Dates: First submitted 2016-04-28; First posted 2016-05-04 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2016-05

CONDITIONS: Undergoing Nonemergent Cardiac Surgery; Central Venous Catheter on the Superior Vena Cava (to Perform ScVO2 Measure); Anemia (<9g/dL) Requiring Blood Transfusion; Hemodynamic and Respiratory Stability; Bleeding Graded as Insignificant, Mild, Moderate of Universal Definition of Perioperative Bleeding
Keywords: Cardiac surgery; Blood transfusion; ScvO2
MeSH Terms: conditions — Anemia; Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ScVO2 group (Experimental): Anemia (<9g/dL) requiring blood transfusion Measure of ScvO2 : ScVO2 is measured using the central venous catheter placed in the superior vena cava. Transfusion is performed if the ScVO2 is inferior or equal to 65%.
  Interventions: Other: ScvO2 measure
- Control group (Other): Anemia (<9g/dL) requiring blood transfusion : Transfusion is performed following national guidelines for red blood cell transfusion
  Interventions: Other: Red blood cell tranfusion

INTERVENTIONS:
Other: Red blood cell tranfusion — Red blood cell transfusion according to transfusion guidelines.
  Arms: Control group
Other: ScvO2 measure — ScvO2 (oximetry) is measured at the distal lumen of the central venous catheter placed in the superior vena cava. Transfusion is performed if ScvO2 is inferior or equal to 65%.
  Arms: ScVO2 group

SUMMARY:
Current international guidelines suggest a restrictive transfusion strategy, setting that Hb level at 7 g/dl is a reasonable threshold. However, the idea of having only one threshold for all the patients has been challenged by authors, suggesting a more liberal strategy for certain cases. At the moment, there is no other parameter considered accurate enough to be taken into consideration for transfusion strategy management.

This study is to use ScVO2, a current, easily accessible parameter, before blood transfusion in order to stratify its indication after cardiac surgery.

Monocentric, randomised, single blind study (patient not aware of the group assignments) Patient inclusion will be made in ICU if the physician decides to perform blood transfusion according to standard transfusion strategy to treat a postoperative anemia (Hb<9g/dL).

Every patient will go through randomization to be placed in one of the two groups of the study: either the one whose transfusion strategy is adjusted by the pretransfusion ScvO2 (group ScvO2), or the control group.

Our main objective is to evaluate the impact of a new transfusion strategy founded on guidelines, but provided ScvO2 is less than 65%, on the incidence of red blood cells transfusion for anemia early after cardiac surgery.

DETAILED DESCRIPTION:
Currently, the rate of transfusion of cardiac surgery patients is approximately 50%. The decision to transfuse is based on the hemoglobin (Hb), the transfusion threshold from 7 to 9 g / dL seems to be reasonable, based on clinical parameters, as well as patient history, as the degree of coronary stenosis . Several randomized studies have shown that a restrictive transfusion strategy was superior to a liberal strategy.

ScvO2 is a parameter reflecting the balance between transport O2 and O2 in tissue consumption, which Hb is one of the determinants. It requires that a levy on central venous used frequently for such patients. ScvO2 could make better account of the actual tolerance of anemia that the only value of Hb and the patient's clinical characteristics.

We therefore hypothesize that ScvO2 can help with the decision of RBC transfusions after heart surgery.

Primary and secondary endpoints Principal: To assess the value of ScvO2 threshold (65%) in the restrictive transfusion strategy on the incidence of transfusion after cardiac surgery.

secondary:

* Assess the impact of transfusion strategy based on ScvO2 on the number of transfused patients at D28
* Assess the impact of transfusion strategy based on ScvO2 on the number of cells transfused concentrates.
* Assess the impact of transfusion strategy based on ScvO2 on mortality or incidence of disease events such as cardiac complications, renal, respiratory or neurological dysfunction in the immediate aftermath of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Patients admitted to intensive care after heart surgery
* Anemic patient (Hb < 9 g/dL)
* Patient with a central venous catheter in the territory SVC

Exclusion Criteria:

* Patient with acute bleeding defined as a postoperative bleeding over 1000 ml in 12 hours or the need for a recovery operation for hemostasis or the transfusion of blood units over 4
* Patient with severe sepsis or septic shock criteria defined by the Surviving Sepsis compaign

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2018-10-17 (Actual)

PRIMARY OUTCOMES:
Number of patients transfused | Between 1 and 28 days (ICU stay)
  Number of patients transfused during ICU stay

SECONDARY OUTCOMES:
Number of patients transfused | Day 28
  Number of patients transfused on day 28
Number of blood units transfused in ICU | Between 1 and 28 days (ICU stay)
  Number of blood units transfused during ICU stay
Number of blood units transfused on day 28 | Day 28
  Number of blood units transfused

OTHER OUTCOMES:
Incidence of mortality | Day 28
  Incidence of 28-day mortality
total duration of mechanical ventilation | Day 1 to 28
  total duration of mechanical ventilation on D28
length of stay in ICU | Day 1 to 28
  The length of stay in ICU
length of hospital stay | Between 1 and 28 days
  The length of stay during hospitalization (Between 1 and 28 days)
Organ failure incidence | Day 1 to 28
  incidence of organ failure at day 28

CONTACTS AND LOCATIONS:
Overall Officials: Norddine ZEOURAL, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- UHMontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided